CLINICAL TRIAL: NCT03369743
Title: Multicentric Data Collection: Virologic Effectiveness at W48 of the Dual Therapy Etravirine (400 mg) + Raltegravir (800 mg) by Once Daily in HIV-positive Patients, Previously Handled by a Dual Etravirine (200 mg x 2/Day) + Raltegravir (400 mg x 2/Day) Taken Twice a Day
Brief Title: Dual Therapy Etravirine + Raltegravir by Once Daily in HIV-positive Patients (ETRAL QD)
Acronym: ETRALQD
Status: Completed | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 007
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Efficacy of etravirin + raltegravir dual therapy was showed in the ANRS 153 ETRAL protocol, in HIV-1 seropositive patients. The use of these two drugs avoids the use of nucleoside reverse transcriptase inhibitors and protease inhibitors, with a real benefit in older patients, who increasingly present contraindications to these drugs' families. The disadvantage of this strategy is twice daily (BID). Pharmacological data suggest that etravirine once a day and raltegravir once a day may provide the same virological efficacy.

The objective of our study is to evaluate the ability of ETRAL QD (etravirine 400 mg x1/day + raltegravir 800 mg x1/day) to maintain virologic success at week 48 (W48), after switch, in HIV-patients under ETRAL BID (etravirine 200 mg x2/day + raltegravir 400 mg x2/day). Virological success is defined as absence of virological failure, and virological failure is defined as two consecutive plasma viral loads >50 cp/ml over 2-4 weeks, or one plasma viral load >400 cp/ml.

This study will be a multicentric data collection. Data will be collected at W0 (patient characteristics, plasma viral load) and then at W4, W12, W24 and W48 (plasma viral load). If stopping strategy, the reason for stopping will be documented. 125 patients will be included in the six participating centers. Data will be centralized at Pitié-Salpêtrière hospital, Paris, with an anonymized e-CRF.

DETAILED DESCRIPTION:
The cART in one taken only a day (QD) improve the quality of life and promote the observance, especially in older patients with cognitive impairment beginning. The ETR+RAL (ETRAL) QD dual therapy should be evaluated.

ETR is a molecule to long half-life (30-40 hours) manageable in QD. SENSE study showed virological efficiency of ETR QD in combination with two NRTIs, and several studies have shown comparable plasma exposure for ETR BID and ETR QD.

The half-life of RAL is shorter (9 hours), but plasma exposure there still seems comparable to RAL BID and RAL QD (same AUC, more important and residual peak lower). Clinical trial of phase III QDMRK also pointed out the non-inferiority of virologic effectiveness of RAL QD compared to RAL BID, in association to two NRTIs, in patients with a pretherapeutic pVL < 100,000 cp/ml.

ODIS clinical trial also showed the effectiveness of RAL QD in combination with two NRTIs (risk of virologic failure increased in case of mutation of prior resistance to the NRTI). The Federal BID to RAL QD switch finally was evaluated in a pilot, to the Pitié-Salpêtrière hospital, all combined cART (tri - and dual therapy), with maintaining a pVL < 50 cp/ml to W48 in 68/71 patients (96%).

Currently, at the Pitié-Salpêtrière hospital, 34 patients on dual therapy ETRAL QD (outside the Protocol), since 137 months median (IQR 41-201), maintain a pVL < 50 cp/ml, suggesting a virologic effectiveness to completely reassuring.

The dual therapy etravirine + raltegravir (ETRAL) in once daily (QD) maintains W48 virological control, switch in patients who were under ETRAL taken twice a day (BID)

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adult
* Treatment by ETRAL BID (etravirine 200 mg x 2/day + raltegravir 400 mg x 2/day) for at least 96 weeks
* plasma Viral Load < 50 cp/ml the day of the switch for ETRAL QD

Exclusion Criteria:

* Virologic failure under ETRAL BID (two consecutive plasma Viral Load < 50 cp/ml)
* Applies contraindicated with etravirine
* Current pregnancy or pregnancy desire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-patients under ETRAL BID (etravirine 200 mg x2/day + raltegravir 400 mg x2/day)
  This study will be a multicentric data collection. Data will be collected at W0 (patient characteristics, plasma viral load) and then at W4, W12, W24 and W48 (plasma viral load)
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Measure of plasma viral load to assess the effectiveness of the dual Etral Qd to maintain the virological success to W48 | 12 months
  Measure ol plasma viral load assessed by RNA quantification using COBAS 6800 system (Roche)

CONTACTS AND LOCATIONS:
Overall Officials: Romain Palich, MD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Yasmine Dudoit, Paris, France

IPD SHARING:
Plan to Share IPD: No